CLINICAL TRIAL: NCT01738282
Title: A Randomized, Multicentric, Double Blind Study to Assess the Efficacy of Xylka® (Baclofen) at the Target Dosage of 180mg/Day Compared to Placebo, for Maintenance of Abstinence in Alcohol Dependent Patients
Brief Title: Efficacy and Safety of Baclofen for Maintenance of Abstinence in Alcohol Dependent Patients
Acronym: ALPADIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethypharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALP 2011007/002
Record Dates: First submitted 2012-11-26; First posted 2012-11-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Alcohol Dependence
Keywords: baclofene; Alcohol dependence; Maintenance of abstinence
MeSH Terms: conditions — Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Experimental): Baclofen 20mg tablet. Titration:increasing dosage regimen to reach the target dosage of 180 mg (9 tablets)in 7 weeks Maintenance period with a constant dosage during 17 weeks Progressive decrease and stop of study treatment in 2 weeks
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Placebo tablet Titration:increasing dosage regimen to reach the target dosage of 9 tablets in 7 weeks Maintenance period with a constant dosage during 17 weeks Progressive decrease and stop of study treatment in 2 weeks
  Interventions: Drug: Placebo (for baclofen)

INTERVENTIONS:
Drug: Baclofen
  Arms: Baclofen
Drug: Placebo (for baclofen)
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy of Xylka® (baclofen) compared to placebo on continuous abstinence rate during 20 weeks of treatment, after withdrawal, in alcohol dependent patients receiving Brenda therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients meeting DSM IV(Diagnosis and Statistical Manual of Mental Disorders, 4th edition) criteria for alcohol dependence
* Willing to participate in the study and express a desire to achieve the objective of continuous and long term abstinence after withdrawal
* Abstinent (last drinking) for a minimum of 3 days and maximum of 14 days
* At least one previous abstinence attempt

Exclusion Criteria:

* Need for a stay at the end of the withdrawal period in a health care and rehabilitation institution specialized in addiction
* Need for a heavy psychosocial out of hospital care
* History of baclofen intake, by prescription or self medication
* Porphyria
* Concomitant treatment with one or several drugs for the maintenance of abstinence
* Severe renal, cardiac or pulmonary disorder
* Epilepsy or history of epilepsy
* Concomitant treatment with psychotropic drugs, except antidepressants at stable dose for 2 months, diazepam and oxazepam
* Severe psychiatric disease (schizophrenia and bipolar disorder)
* Suicidal risk or history of suicide
* Clinically significant cognitive disorders
* Hepatic encephalopathy
* Ongoing dependence or within the last 12 months on other addictive substances (opioid, cocaine, cannabis, other substances or drugs…), excepted tobacco

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence rate in each group (baclofen or placebo) during 20 weeks of treatment, from Day 29 to Day 168. | Day 168

SECONDARY OUTCOMES:
Continuous abstinence rate from the first intake of study treatment (Day 1) to the end of the maintenance dose period (Day 168), i.e. 24 weeks | Day 168
Continuous abstinence rate from the first intake of study treatment (Day 1) to the end of 4-week post treatment follow up period (Day 210), i.e. 30 weeks | Day 210
Continuous abstinence rate during 20 weeks of treatment (Day 29 to Day 168), according to the severity of alcohol dependence | Day 168
Continuous abstinence rate during 20 weeks of treatment (Day 29 to Day 168), according to the level of drinking before withdrawal (Time Line Follow Back calendar/ World Health Organization criteria for risk of consumption) | Day 168
Drinking characteristics for patients having a relapse between Day 1 and Day 210 | Day 210
  Time to relapse (Day 1 to first drinking day) Time to relapse to first high risk drinking day (>60g for a male, > 40g for a female) Percentage of drinking days from Day 1 to Day 210 Mean number of standard drinks per drinking day and classification according to World Health Organization criteria for the risk of consumption Percentage of high risk drinking days during the maintenance period at the target dosage (Day 50 to Day 168) compared to the percentage of high risk drinking days during the preceding 4 weeks of the withdrawal Percentage of drinking days during the maintenance period at the target dosage (Day 50 to Day 168) compared to the percentage of drinking days during the preceding 4 weeks of the withdrawal
Change in craving, addiction and Quality of Life scales | Day 210
  Clinical Global Impression (CGI), Alcohol dependence Quality of Life (AlQoL9), Obsessive Compulsive Drinking Scale (OCDS), Hospital Anxiety and Depression Scale (HAD), Visual Analogue Scale (VAS) craving scores and liver biomarkers
Recording of safety data | Day 210
  Adverse events, vital signs, biological parameters, ECG and urinary pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Michel REYNAUD, MD, Principal Investigator — Villejuif, France
Locations (38):
- France (38):
  - Angers
  - Bron
  - Clermont de l'Oise
  - CHU, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Dax
  - Centre hospitalier, Dijon
  - Centre hospitalier, Erstein
  - Centre hospitalier, La Membrolle-sur-Choisille
  - Hopital Michallon, La Tronche
  - LArbresle
  - Centre hospitalier, Le Mans
  - CHRU, Lille
  - CSAPA, Lille
  - Limoges
  - Hopital de la Croix Rousse, Lyon
  - Hopital Sainte Marguerite, Marseille
  - Centre hospitalier, Montauban
  - Morlaix
  - Hopital Villemin, Nancy
  - CHU, Nantes
  - Centre hospitalier, Nice
  - CHRU, Nîmes
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Cochin, Paris
  - Hopital Fernand Widal, Paris
  - Hopital Saint Anne, Paris
  - Centre hospitalier, Perpignan
  - Centre hospitalier, Pont-du-Casse
  - Reims
  - Hopital Pontchaillou, Rennes
  - Hopital de la Fraternité, Roubaix
  - Saint-Égrève
  - Hopital René Muret, Sevran
  - CSAPA, Seynod
  - Centre hospitalier intercommunal, Toulon
  - Hopital Brabois, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif

REFERENCES:
- [Derived] Braillon A, Naudet F. Pharmacotherapies for Alcohol Use Disorder: Over Both Sides of the Atlantic Ocean. Mayo Clin Proc. 2020 Oct;95(10):2294-2295. doi: 10.1016/j.mayocp.2020.08.005. No abstract available. PMID 33012365